## **Informed Consent Form**

TITLE: Biomarkers for Event-driven PrEP Adherence

**NCT NUMBER:** NCT04298697

**IRB APPROVAL DATE:** December 1, 2021

## You Are Being Asked to Be in a Research Study ARM B

You are being asked to be in a research study. A research study is designed to answer a scientific question. If you agree to be in the study you will be one of 40 people who are being studied, at Emory University Hope Clinic.

## Why is this study being done?

This study is being done to answer the question: How useful are biomarkers to confirm self-reported adherence to event-driven PrEP. You are being asked to be in this research study because you identify as a man who has sex with men and you are between the ages of 18 and 59 years old.

## Do you have to be in the study?

It is your decision to be part of this research study. You do not have to be in it. Your choice will not affect your access to medical care. Before you make your decision, you should take time to learn about the study.

## What do I have to do if I choose to participate in this study?

If you are eligible and want to be part of the study, you will participate for no more than 24 weeks (21 study visits). The researchers will ask to collect the following samples from you: blood, hair, urine, and a finger stick.

## What are the risks or discomforts I should know about before making a decision?

The drug provided in this study will not protect participants from HIV or treat any active HIV infections. All studies have some risks. Some risks are relatively small, like being bored or losing time. Some are more serious – for this study, the drugs that are tested have been shown to be well tolerated, but can include common side effects such as, diarrhea, nausea, and headaches. Tenofovir and emitricitabine (TDF/FTC) can also cause flare-ups in those who have hepatitis B virus. The risks of loss of privacy and breach of confidentiality are rare but can occur. A full list of expected risks, their frequency and severity are in the "What are the possible risks and discomforts?" section of this document.

#### Alternatives to Joining This Study

Since this is not a treatment study, the alternative is not to participate or to consider participating in another study.

#### Costs

You WILL NOT have to pay for any of the study procedures while participating in this study. There is more information in the cost section below.

#### What Should I Do Next?

Read this form, or have it read to you. Make sure the study doctor or study staff explains the study to you. Ask questions (e.g., about exact time commitment, about unfamiliar words, more details on specific procedures, etc.). Take time to consider this and talk about it with your family and friends.

Version Date: 08/16/2021

# Emory University Consent to be a Research Subject – Arm B

Title: Biomarkers for Event-Driven PrEP Adherence

Principal Investigator: Colleen F. Kelley MD, MPH

**<u>Study-Supporter:</u>** Center for Disease Control and Prevention (CDC)

#### Introduction

You are being asked to be in a medical research study. This form is designed to tell you everything you need to think about before you decide if you want to be a part of the study. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the research study. The decision to join or not join the research study will not cause you to lose any medical benefits. If you decide not to take part in this study, your doctor will continue to treat you.

Before making your decision:

- Please carefully read this form or have it read to you
- Please listen to the study doctor or study staff explain the study to you
- Please ask questions about anything that is not clear

You can take a copy of this consent form, to keep. Feel free to take your time thinking about whether you would like to participate. You may wish to discuss your decision with family or friends. Do not sign this consent form unless you have had a chance to ask questions and get answers that make sense to you. By signing this form, you will not give up any legal rights.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## What is the purpose of this study?

The purpose of this study is to understand how useful biomarkers are to confirm self-reported adherence to event-driven PrEP in men who have sex with men. The study drug being examined in this study is Truvada. The study drug provided is not intended to protect you from HIV or treat any active infection.

This study will consist of 40 healthy, HIV-negative men, aged 18-59, who have sex with men. There are a total of 4 arms in this study (A, B, C, & D.) You are being asked to participate in Arm B. There will be a total of 20 men in this study arm. Study participants will take 2-1-1 dosing of the study drug. This means you will take 2 pills first, then 1 pill 24 hours later, then another pill 48 hours later. The researchers will then take biological samples from participants and measure the amount of drug in the samples. Biological samples that will be taken include blood, hair, urine, and a finger stick.

#### What will I be asked to do?

If you decide to take part in this study, you will be asked to come to the Hope Clinic to complete 21 visits over a period of 24 weeks.

**Visit 1 (Screening):** If you agree to be in the study, this visit will likely take place on the same day you sign the consent form. The purpose of this visit is to see if you are a good fit for the study. During this visit, you will be asked questions about your medical and sexual history and have an HIV blood test done. You may also undergo a physical exam. Before and after HIV testing, we will counsel you about the test and results. We will draw approximately 24 mL of blood (about 3 teaspoons) from your arm for other blood tests to see if you have

Version Date: 08/16/2021

hepatitis B and to see whether your kidney function is normal. If you are eligible to take part in the study, we will schedule you for your second study visit 1-6 weeks after your first visit.

**Visit 2 (Enrollment):** At this visit we will give you your first dose of the study drug (2 pills.) You will take the first dose of 2 pills while you are still in the clinic. At this visit you will also be given the next dose to be taken 24 hours later, as well as the dose to take 48 hours later. In addition to that, you will be given your weekly 2-1-1 doses for the next 2 weeks to be taken at home. Since you will take these doses on your own, we will ask you to take a time stamped photograph or videotape of yourself taking the pill. You will also have the option to send a text to a specified number with the time and date of dose if your phone device does not have video/photo capabilities. These doses will need to be taken weekly, on the same days every week.

## **Types of Samples**

## Standard Biological Samples

There are a set of biological samples that will be collected from all participants at each post-dose visit (Visits 3-21). We will refer to them as "standard samples" for the rest of this document. The standard samples include:

- Blood: We will draw approximately 24 mL (about 5 teaspoons) of blood from your arm.
- Urine sample: Some of which will be used for gonorrhea and chlamydia testing.

## Hair Sample

At visits 6, 10, 14 and 21 (monthly) we will also ask for:

• Hair sample: we will cut a small sample (about 50-100 strands) with scissors.

The timing of the visits is very important in this study so it is important that you keep all scheduled appointments.

#### Visit 3

This visit will begin your weekly convenience sampling. You will need to come to the clinic at any point during the week for us to take the standard samples.

## Visit 4

You will need to come to the clinic at any point during the week for us to take the standard samples.

#### Visit 5

You will need to come to the clinic at any point during the week for us to take the standard samples. We will also give you your next supply of the study drug at this visit.

#### Visit 6

You will need to come to the clinic at any point during the week for us to take the standard samples plus a hair sample. We will also complete an HIV test at this visit.

## Visit 7

You will need to come to the clinic at any point during the week for us to take the standard samples.

#### Visit 8

You will need to come to the clinic at any point during the week for us to take the standard samples. We will also give you your next supply of the study drug at this visit.

#### Visit 9

You will need to come to the clinic at any point during the week for us to take the standard samples.



## Visit 10

You will need to come to the clinic at any point during the week for us to take the standard samples plus optional hair samples. We will also complete a rapid HIV test as well as rectal and urine STI screening at this visit.

#### Visit 11

You will need to come to the clinic at any point during the week for us to take the standard samples. We will also give you your next supply of the study drug at this visit.

#### Visit 12

You will need to come to the clinic at any point during the week for us to take the standard samples.

#### Visit 13

You will need to come to the clinic at any point during the week for us to take the standard samples.

## Visit 14

You will need to come to the clinic at any point during the week for us to take the standard samples plus an optional hair sample. At this visit we will also do an HIV test and a creatinine test.

#### Visit 15

You will take your final 1 pill dose in clinic before we take standard samples.

#### Visit 16

For this visit, you will need to come into the clinic 24 hours after your last dose at Visit 15. Standard samples will be taken.

#### Visit 17

For this visit, you will need to come into the clinic 2-5 days after your last dose at Visit 15. Standard samples will be taken.

#### Visit 18

For this visit, you will need to come into the clinic 7 days after your last dose at Visit 15. Standard samples will be taken.

#### Visit 19

For this visit, you will need to come into the clinic 14 days after your last dose at Visit 15. Standard samples will be taken.

#### Visit 20

For this visit, you will need to come into the clinic 21 days after your last dose at Visit 15. Standard samples will be taken.

#### Visit 21

For this visit, you will need to come into the clinic 28 days after your last dose at Visit 15. Standard samples will be taken plus a hair sample.

As a participant in a Hope Clinic study, your overall health is important to us. Because the treatment regimen outlined in this document is not approved to prevent HIV, if you feel at any point during your participation on this study that you may have been exposed to HIV, we will refer you to a healthcare provider who can provide Post-exposure Prophylaxis (PEP).

Version Date: 08/16/2021



## How will my medicine be provided?

The medicine that you will take will be dispensed by the pharmacy and delivered to the principal investigator or study team member. The principal investigator or health care providers on his/her research team will provide the medicine to you. If you have questions about the medicine, you should ask the principal investigator or study nurse. You may also call the pharmacy at the pharmacy at the pharmacy is included on your medicine package.

#### Who owns my study information and samples?

If you join this study, you will be donating your samples and study information. You will not receive any compensation if your samples or information are used to make a new product. If you withdraw from the study, data and samples that were already collected may still be used for this study. If you decide to withdraw from the study and would like us to destroy any remaining sample, please contact Dr. Kelley in writing at:



## What are the possible risks and discomforts?

There may be side effects from the study drug or procedures that are not known at this time. Everyone taking part in the study will be watched carefully for any side effects. Most side effects go away soon after stopping Truvada. You should talk to the study doctor about any side effects that you experience while taking part in this study.

Possible risks and discomforts related to the study procedures include the following:

## STI Testing

It is possible that you will find out that you have HIV, gonorrhea or chlamydia during this study. This could cause you some stress. Study staff will be available for counseling before and after your test, regardless of the results. Also, we will refer you to a medical provider for further care.

#### **Blood Draw**

Having your blood taken can cause discomfort. This discomfort is temporary but may cause lightheadedness or fainting. Taking blood can cause bruising. Bruising can be prevented or reduced by putting pressure on the site for a few minutes after the blood is taken. Rarely, some people get an infection where the needle was put in their arm to draw the blood. To reduce the risk of infection, we will wipe the area clean with alcohol and use sterile equipment.

## Truvada (TDF/FTC)

Truvada (TDF/FTC) is a combination anti-HIV medication that contains the drugs tenofovir and emtricitabine. Based on clinical trials previously conducted of TDF/FTC, the drug showed to be well tolerated (see package insert). The most common adverse events reported in clinical trials ( $\geq$  5% incidence) included diarrhea, nausea, and headache. Additional adverse reactions occurring in less than 2% of subjects administered TDF/FTC included vomiting, flatulence, dyspepsia, abdominal pain, rash, and depression.

Renal toxicity and bone density loss are rarely reported with chronic use of TDF containing products and are not expected to occur with the regimen prescribed in this protocol. Similarly, lactic acidosis and severe hepatomegaly have rarely been associated with medications in the same class as TDF and FTC.

Version Date: 08/16/2021

Use of TDF/FTC can also cause flare-ups in those who have hepatitis B virus. It can cause the Hepatitis B virus to suddenly return in a worse form than before if treatment was provided (see package insert). For this reason, it is important that participants not participate in the study if they are known to have Hepatitis B.

If you will be taking the study drug home, keep it out of the reach of children or anyone else who may not be able to read or understand the label. Do not let anyone else take the study drug besides you.

The medication provided in this study is not for treatment or prevention of HIV infection, and you should not expect that you will be protected from HIV by taking the medications in this study. If you are interested in pre-exposure prophylaxis (PrEP) after this study ends, we can refer you to a medical provider who can prescribe PrEP.

#### **New Information**

It is possible that the researchers will learn something new during the study about the risks of being in it. If this happens, they will tell you about it. Then you can decide if you want to continue to be in this study or not. You may be asked to sign a new consent form that includes the new information if you decide to stay in the study.

## Will I benefit directly from the study?

This study is not designed to benefit you directly. This study is designed to evaluate the usefulness of biomarkers to confirm self-reported adherence to event-driven PrEP. The study results may be used to help others in the future if this regimen is one day an approved pre- exposure prophylaxis (PrEP) regimen.

## Will I be compensated for my time and effort?

Compensation will be provided on a web based, reloadable, debit card (ClinCard) that automates reimbursements. The ClinCard will be provided by study staff at the initial visit (visit 1).

All payments are made using a personal payment card. We issue this to you for free. The payment card is a prepaid debit card. It can be used exactly like a MasterCard. We load money onto your card electronically every time you need to be paid. The card scheme is run by Greenphire, an independent company specializing in payments for research studies and clinical trials. To issue your card, we need to give Greenphire some of your personal information. Banks and other financial institutions can access this information if they need to verify your identity when you use your card.

Emory University is required by law to report any payments we make to the IRS. To do this, Emory University Department of Finance needs to keep your Social Security Number on file. We are asking you to allow us to communicate your name, address, date of birth, research study name and Social Security Number to Greenphire and Emory University Department of Finance. If you want to receive e-mail or text alerts when payments are made to you, we will ask you to provide your e-mail or phone number as well. All of this information will be stored on computers owned by Greenphire. Greenphire will not have access to any other information collected during this study. Full instructions about using your card are included when we issue it. Please ask if you have any questions or concerns about the card scheme.

We would also like the option of compensating you in the form of cash, check or gift card if ClinCard accessibility is not available. You may be asked to fill out a tax form, including your Social Security or Taxpayer Identification Number, in order to be reimbursed, depending on the amount and method of payment. Some payment methods involve mail coming to your house, which may be seen by others in your household. You can decline payment if you are concerned about confidentiality, or you can talk to the study team to see if there are other payment options.

You will get \$50 for each visit to compensate you for your time and effort. If you do not finish the study, we will compensate you for the visits you have completed. You will get \$1050 total, if you complete all study visits. We

permit missing up to three visits (completing 18 visits.) If you complete 18 visits for the study, you will receive a \$100 bonus for completion of the study, for a total of \$1150. If an extra study visit is necessary, you will receive \$20 for completion of that study visit.

If you have trouble with transportation to study visits, please let the study staff know. We may be able to help (e.g. MARTA ride card).

#### What are my other options?

If you decide not to enter this study, there is care available to you outside of this research study. The study doctor will discuss these with you.

Taking part in this study, however, may make you unable to participate in some other research studies, if they exclude people who have taken certain treatments. You should discuss this with the researchers if you have concerns. You may wish to research other study options at websites like clinicaltrials.gov and ResearchMatch.org.

## How will you protect my private information that you collect in this study?

Whenever possible, a study number, rather than your name, will be used on study records. Your name and other identifying information will not appear when we present or publish the study results.

Certain offices and people other than the researchers may look at study records. Government agencies and Emory employees overseeing proper study conduct may look at your study records. These offices include the Food and Drug Administration (FDA), the Office for Human Research Protections, the sponsor, the Emory Institutional Review Board, the Emory Office of Research Compliance. Study funders may also look at your study records. Emory will keep any research records we create private to the extent we are required to do so by law. A study number rather than your name will be used on study records wherever possible. Your name and other facts that might point to you will not appear when we present this study or publish its results.

#### **Certificate of Confidentiality**

There is a Certificate of Confidentiality from the National Institutes of Health for this Study. The Certificate of Confidentiality helps us to keep others from learning that you participated in this study. Emory will rely on the Certificate of Confidentiality to refuse to give out study information that identifies you. For example, if Emory received a subpoena for study records, it would not give out information that identifies you.

The Certificate of Confidentiality does not stop you or someone else, like a member of your family, from giving out information about your participation in this study. For example, if you let your insurance company know that you are in this study, and you agree to give the insurance company research information, then the investigator cannot use the Certificate to withhold this information. This means you and your family also need to protect your own privacy.

The Certificate does not stop Emory from making the following disclosures about you:

- Giving state public health officials information about certain infectious diseases,
- Giving law officials information about abuse of a child, elderly person or disabled person.
- Giving out information to prevent harm to you or others.

Giving the study sponsor or funders information about the study, including information for an audit or evaluation.

#### Storing and Sharing your Information

Samples collected during the study will be sent to the Centers for Disease Control (CDC) for testing.

De-identified data from this study (data that has been stripped of all information that can identify you), including your de-identified genetic information, may be placed into public databases where, in addition to having no direct identifiers, researchers will need to sign data use agreements before accessing the data. We will remove or code any personal information that could identify you before your information is shared. This will ensure that, by current scientific standards and known methods, it is extremely unlikely that anyone would be able to identify you from the information we share. Despite these measures, we cannot guarantee anonymity of your personal data.

Your data and specimens from this study may be useful for other research being done by investigators at Emory or elsewhere. To help further science, we may provide your de-identified data and/or specimens to other researchers. If we do, we will not include any information that could identify you. If your data or specimens are labeled with your study ID, we will not allow the other investigators to link that ID to your identifiable information.

We will use your sample and data only for research. We will not sell them. However, the results of this research might someday lead to the development of products (such as a commercial cell line, a medical or genetic test, a drug, or other commercial product) that could be sold by a company. You will not receive money from the sale of any such product.

In general, we will not give you any individual results from the study of the samples you give us. If we find something of urgent medical importance to you, we will inform you, although we expect that this will be a very rare occurrence.

#### **Future use of specimens**

Leftover specimens may be stored for future research use at the CDC or at the Hope Clinic. You cannot participate in this protocol if you do not want your specimens stored for possible future use. At this time, there are no plans for genetic testing of the specimens. However, it is possible that researchers may choose to do genetic testing in the future on the stored specimens. Your name and personal identifying information will not be labeled on the stored specimens.

## How is my Genetic Information Protected? What are the Risks?

The Genetic Information Nondiscrimination Act (GINA) is a federal law that generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when making a decision to hire, promote, or fire you or when setting the terms of your employment.

Be aware that GINA does <u>not</u> protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance, and does not apply to employers with less than 15 employees.

In addition to GINA, the State of Georgia has laws that prohibit insurers from using genetic testing information for any non-treatment purpose. However, like GINA, this state law protection has exclusions: life insurance policies, disability income policies, accidental death or dismemberment policies, Medicare supplement policies, long-term care insurance policies, credit insurance policies, specified disease policies, hospital indemnity

Version Date: 08/16/2021

policies, blanket accident and sickness policies, franchise policies issued on an insurance policy written as a part of workers' compensation equivalent coverage, or other similar limited accident and sickness policies.

## Privilege

In the State of Georgia, in some circumstances your genetic information may have special legal protections called "privilege." This means that the information cannot be used as evidence in a court. By allowing us to use and disclose your genetic information for this research study along with other information about you that genetic information used in the research may no longer have that legal protection. Other protections described in this form will still apply. There are also other confidentiality protections for research data in general under Georgia state law.

## Storage and release of samples, genomic data, and health information

Portions of your samples, genomic data, and health information will be stored and shared with other researchers. The samples and information will be available for any research question, such as research to understand what causes certain diseases (for example heart disease, cancer, or psychiatric disorders), development of new scientific methods, or the study of where different groups of people may have come from.

## **Unrestricted access databases**

If researchers choose to do genetic testing in the future on stored specimens, the information from this study will be freely available in a public, unrestricted database that anyone can use. The public database will include information on hundreds of thousands of genetic variations in your DNA code, as well as your ethnic group and sex. The only health information included will be whether you had a particular disease or not. This public information will not be labeled with your name or other information that could be used to easily identify you. However, it is possible that the information from your genome, when combined with information from other public sources could be used to identify you, though we believe it is unlikely that this will happen.

## **Medical Record**

If you have been an Emory Healthcare patient before, then you already have an Emory Healthcare medical record. If you have never been an Emory Healthcare patient, you do not have one. An Emory Healthcare medical record will be made for you if an Emory provider or facility gives you any services or procedures for this study.

We will take reasonable steps to keep copies of this form out of Emory Healthcare's medical records system. If we aren't successful in keeping these forms out, despite our efforts, we will take steps to remove them. If they cannot be removed, we will take steps to limit access to them.

Emory Healthcare may create study information about you that can help with your care. For example, the results of study tests or procedures. These study results will be put in your Emory Healthcare medical record. Anyone who has access to your medical records will be able to have access to all the study information placed there. The confidentiality of the study information in your medical record will be protected by laws like the HIPAA privacy rule. State and federal laws may not protect the research information from disclosure. We will ask for your authorization if we need to obtain any information from your medical record.

We will also keep a separate research record of all study tests and procedures that we will use for research purposes. This research record will not be a part of your medical record. For this study, those items include:

- Medical History & Physical Examination
- Laboratory testing
- HIV testing & Pretest Counseling

Tests and procedures done at non-Emory places may not become part of your Emory medical record. Also, if you decide to be in this study, it is up to you to let your other health providers know.



## **Return of research results**

Except for your HIV and STI test results, we will not give you any individual results from the study of the samples you give us. If we find something of urgent medical importance to you, we will inform you, although we expect that this will be a very rare occurrence.

## In Case of Injury

If you believe you have become ill or injured from this research, you should contact Dr. Colleen Kelley at telephone number . You should also let any health care provider who treats you know that you are in a research study.

If you get ill or injured from being in the study, Emory will help you to get medical treatment. Neither Emory nor the sponsor will pay for your medical treatment. Your insurer will be billed for your treatment costs. If you do not have insurance, or if your insurance does not pay, then you will have to pay these costs.

Emory and the sponsor have not, however, set aside any money to pay you if you are injured as a result of being in this study or to pay for this medical treatment. For Emory, the only exception is if it is proven that your injury or illness is directly caused by the negligence of an Emory employee. "Negligence" is the failure to follow a standard duty of care. You do not give up any legal rights you may have by being in this study, including any right to bring a claim for negligence.

#### Costs

There will be no costs to you for participating in this study, other than basic expenses like transportation. You will not be charged for any of the research activities. If the study procedures result in any medical complications that would not fall under "injury" as discussed above, the cost of treatment for those complications may be charged to you or your insurance.

## Withdrawal from the Study

You have the right to leave a study at any time without penalty.

For your safety, however, you should consider the study doctor's advice about how to go off the study treatment. If you leave the study before the final planned study visit, the researchers may still use your samples unless you revoke your authorization.

The researchers also have the right to stop your participation in this study without your consent for any reason, especially if they believe it is in your best interest or if you were to object to any future changes that may be made in the study plan.

These are the expected reasons why the researchers may stop your participation:

- If you are unable or unwilling to follow all of the study procedures or instructions,
- You could be harmed by study drug and/or study procedures,
- You are not able to attend clinic visits or complete all of the study procedures, or
- Other reasons, as decided by the study staff.

## **Contact Information**

Contact Colleen Kelley MD, MPH at

- if you have any questions about this study or your part in it,
- if you feel you have had a research-related injury or a bad reaction to the study drug, or
- if you have guestions, concerns or complaints about the research

For emergency use only, 24 hr. pager:



Contact the Emory Institutional Review Board at 404-712-0720 or 877-503-9797 or irb@emory.edu:

- if you have questions about your rights as a research participant.
- if you have questions, concerns or complaints about the research.
- You may also let the IRB know about your experience as a research participant through our Research Participant Survey at <a href="http://www.surveymonkey.com/s/6ZDMW75">http://www.surveymonkey.com/s/6ZDMW75</a>.

## **Consent**

## Optional Videotape or Photograph You At-Home Drug Dose:

You will be asked to videotape or photograph yourself taking your weekly doses of Truvada at home with your smart phone. We ask you to do this so we can verify when you took the study drug. Your other option would be to text a designated phone number when you take the at-home dose. You will be required to do one or the other in order to participate in the study.

| Your decision to videotape or photograph your dose will not affect your p Please place your initials below (select only ONE option): | articipation i | n this study. |
|---|---|---|
| YES, I agree to videotape or photograph my dose (Initials) | | |
| NO, I do not agree to videotape or photograph my dose | | |
| TO BE FILLED OUT BY SUBJECT O Please print your name, sign, and date below if you agree to be in this r and authorization form, you will not give up any of your legal rights. We will keep. | esearch stu | |
| Name of Subject | | |
| Signature of Subject (18 or older and able to consent) | Date | :am / pm<br>Time |
| TO BE FILLED OUT BY STUDY TEAM | ONLY | |
| Name of Person Conducting Informed Consent Discussion | - | |
| Signature of Person Conducting Informed Consent Discussion | Date | :am / pm<br>Time |

Version Date: 08/16/2021 IRB Form 12142018